CLINICAL TRIAL: NCT02433977
Title: A Proof of Concept Study to Determine the Effects of NOX and Conjugated Linoleic Acid on Asthmatics
Brief Title: The Effects of NOx and Conjugated Linoleic Acid on Asthmatics
Acronym: NICLA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gladwin, Mark, MD (Individual)
Responsible Party: Principal Investigator, Sally E. Wenzel MD, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO14110207
Record Dates: First submitted 2014-12-11; First posted 2015-05-05 (Estimated); Results first posted 2021-03-26 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Asthma
Keywords: Asthma; Obesity; conjugated linolenic acid; nitrate; nitrite; nutritional supplements
MeSH Terms: conditions — Asthma; Obesity | interventions — eleostearic acid; Sodium Nitrite; sodium nitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Conjugated Linolenic Acid + NOx (Experimental): This is a single arm study
  Conjugated Linolenic Acid (CLA)- daily oral dose 3 g/day
  Sodium Nitrate- Capsules for daily oral administration at the dose of 1 g (2 x 500 mg)
  Sodium Nitrite- Capsules for daily oral administration at the dose of 20 mg (2 x 10 mg)
  Interventions: Dietary Supplement: Conjugated Linolenic Acid; Drug: Sodium Nitrite; Drug: Sodium Nitrate

INTERVENTIONS:
Dietary Supplement: Conjugated Linolenic Acid — CLA is a polyunsaturated fatty acid Subjects will receive capsules for daily oral administration at the dose of 3 g/day
  Other Names: conjugated linolenic acid (CLA)
Drug: Sodium Nitrite — Subjects will receive capsules for daily oral administration at the dose of 20 mg (2 x 10 mg)
Drug: Sodium Nitrate — Subjects will receive capsules for daily oral administration at the dose of 1g (2 x 500 mg)

SUMMARY:
This study will examine the hypothesis that in obese asthmatics; treatment with NOx + CLA is well tolerated, safe and will increase eNO while reducing airway oxidative stress. Allied with this, the investigators will define whether supplementing with this bioactive mediator modifies the airway microbiome, and reduces airway inflammation.

DETAILED DESCRIPTION:
Obesity is an asthma comorbidity associated with increased severity, poor control, reduced steroid responsiveness and greater exacerbation and healthcare utilization rates. These associations are not explained by having a greater degree of Th-2 inflammation. Rather, the obese asthma phenotype defined in several cluster studies, has paradoxically reduced levels of Th-2 biomarkers, including sputum eosinophils and exhaled nitric oxide (NO). The investigators previous research has shown that the inverse relation between increased body mass index (BMI) and reduced exhaled NO, may be explained by a metabolic imbalance characterized by lower L-arginine and greater asymmetric di-methyl arginine (ADMA) levels. Having a low L-arginine/ADMA ratio has been shown to inhibit and uncouple all isoforms of nitric oxidase synthase (NOS), thereby reducing NO bioavailability and promoting oxidative stress through enhanced superoxide production. In obese asthmatics, this imbalance not only correlates with exhaled NO, but also with lower FEV1% and poorer asthma-related quality of life. Yet the effect of obesity in asthma is unlikely to be solely dependent on a single mechanism. Other factors, such as increased Th1 and Th-17-mediated inflammation have been shown to occur in human and animal models. Given all of these potential avenues, it is imperative that an intervention is sufficiently pleiotropic that can, in addition to restoring airway NO levels, also reduce other obesity-related non-Th2 mechanism of inflammation. The investigators hypothesize that treatment with conjugated linolenic acid (CLA) + nitrate and nitrite (together known as NOx), will restore NO airway bioavailability, reduce oxidative stress and improve airway inflammation in obese asthmatics. To test this hypothesis, the investigators propose a phase II pilot study in which obese asthmatics with metabolic syndrome, will be treated orally with CLA+NOx for 8 weeks, in an open label study design to assess pre to post-intervention changes in airway and systemic biomarkers, and to determine the effects on lung function and bronchial hyperresponsiveness. Participants will undergo a pre and post intervention bronchoscopy. The results obtained from this project will be greatly informative to our understanding of the obese - asthma pathophysiology and for the development of clinical trials to determine the potential benefit of this intervention in improving health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adequate completion of informed consent process with written documentation
* Male and female patients, ≥ 18 - 65 yrs old
* Diagnosis of asthma: based on previous physician diagnosis and either baseline pre-bronchodilator FEV1 50% or greater predicted with a 12% or greater bronchodilator response to 4 puffs of albuterol or PC20 methacholine (16 mg) if no BD response.If the subject is not currently on an ICS/ ICS LABA, PC20 should be < 8 mg, if no BD response. Spirometry results within the prior 24 months located in the subject's medical records can be used to determine eligibility, if available.
* All racial/ethnic backgrounds with a diagnosis of asthma for ≥6 months
* Smoking history ≤10 pack years and no smoking in the last year
* BMI ≥ 30
* If subject is on ICS or ICS/LABA therapy- 30 days on a stable dose (up to 1,000 mcg daily fluticasone equivalent)
* Asthma diagnosed at age 9 or later

Exclusion Criteria:

* Respiratory tract infection within the last 4 weeks
* Oral or systemic CS burst within the last 4 weeks
* Asthma-related hospitalization within the last 2 months
* Asthma-related ER visit within the previous 4 weeks
* Significant or uncontrolled concomitant medical illness including (but not limited to) heart disease, cancer, diabetes
* Chronic renal failure (creatinine > 2.0) at screening (Associated with higher ADMA levels)
* Current statins use (statins lower ADMA levels), patients may stop and re-enroll after 2 weeks of stopping statins
* Positive pregnancy test
* Intolerance or allergy to the intervention drugs
* Current or recent (within 30 days) in an investigational treatment study.
* Unable or unlikely to complete study assessments or the study intervention (i.e. bronchoscopy) poses undue risk to patient in the opinion of the Investigator.
* Any kind of oral nitrates such as nitroglycerin or already taking supplements
* History of ICU admission/intubation due to asthma in the past year;
* More than three systemic corticosteroid requiring asthma exacerbations in the past year
* Systemic steroid dependent asthma (no daily oral steroids- short term therapy for asthma exacerbation is permitted)
* Use of mouthwash containing chlorhexidine (lowers NO) within 1 week prior to screening and throughout the study
* Untreated sleep apnea
* Hgb A1C ≥7
* Daily use of PPI's (Proton Pump Inhibitor) or H2 Blockers for GERD (it is permitted to take on an occasional basis- no more than 1x per week. If participants wash out of these meds for 1 week, they can enroll)
* Use of biologics for asthma/allergies unless there is a 4 month washout prior to enrollment (the washout for biologics is done for clinical reasons and not specifically for inclusion for the study).
* Drug and/or alcohol abuse for ≥1 year
* Breastfeeding
* Any other condition and/or situation that causes the investigator to deem a subject unsuitable for the study (e.g. due to expected study medication non-compliance, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study-related procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sally E Wenzel, MD, Principal Investigator — The University of Pittsburgh Asthma Institute at UPMC
Locations (1):
- The University of Pittsburgh Asthma Institute at UPMC, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Conjugated Linolenic Acid + NOx: This is a single arm study
  Conjugated Linolenic Acid (CLA)- daily oral dose 3 g/day
  Sodium Nitrate- Capsules for daily oral administration at the dose of 1 g (2 x 500 mg)
  Sodium Nitrite- Capsules for daily oral administration at the dose of 20 mg (2 x 10 mg)
  Conjugated Linolenic Acid: CLA is a polyunsaturated fatty acid Subjects will receive capsules for daily oral administration at the dose of 3 g/day
  Sodium Nitrite: Subjects will receive capsules for daily oral administration at the dose of 20 mg (2 x 10 mg)
  Sodium Nitrate: Subjects will receive capsules for daily oral administration at the dose of 1g (2 x 500 mg)
Period: Overall Study
Arm/Group | Conjugated Linolenic Acid + NOx
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Conjugated Linolenic Acid + NOx
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Exhaled NO Before and After Treatment
Description: Determine how CLA and NOx affect airway NO bioavailability (exhaled NO)
Time Frame: Before treatment at baseline and after treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: parts per billion
Arm/Group | Conjugated Linolenic Acid + NOx
Number analyzed (Participants) | 6
parts per billion | 39.5 (10.4)
Statistical Analysis 1: Comparison: Conjugated Linolenic Acid + NOx; Test type: Other; p <= 0.05, t-test, 1 sided

2. Secondary Outcome: Biomarkers of Inflammation-bronchial Hyperresponsiveness Using PC20
Description: To determine whether, compared to baseline, treatment with NOx + CLA can reduce bronchial hyperresponsiveness. PC20 was measured by methacholine challenge (mg/mL) in three participants pre and post supplementation with Nitrate/Nitrite and cLA
Time Frame: Before treatment at baseline and after treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Conjugated Linolenic Acid + NOx
Number analyzed (Participants) | 3
mg/mL | 10.33 (12.74)
Statistical Analysis 1: Comparison: Conjugated Linolenic Acid + NOx; Test type: Other; p <= 0.05, t-test, 1 sided

3. Secondary Outcome: Biomarkers of Inflammation- Concentration of Free CLA in Plasma
Description: To determine whether, compared to baseline, treatment with NOx + CLA can quantify the concentrations of free CLA in plasma
Time Frame: Before treatment at baseline and after treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: Nanomolar
Arm/Group | Conjugated Linolenic Acid + NOx
Number analyzed (Participants) | 6
Nanomolar | 161.8 (44.3)
Statistical Analysis 1: Comparison: Conjugated Linolenic Acid + NOx; Test type: Other; p <= 0.05, t-test, 1 sided

4. Secondary Outcome: Number of Participants With an Increase in IL-6 and IL-1b Expression
Description: To determine whether, compared to baseline, treatment with NOx + CLA will increase a participant's IL-6 and IL-1b expression.
Time Frame: Before treatment at baseline and after treatment at 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Conjugated Linolenic Acid + NOx
Number analyzed (Participants) | 6
Participants | 5
Statistical Analysis 1: Comparison: Conjugated Linolenic Acid + NOx; Test type: Other; p <= 0.05, t-test, 1 sided

5. Secondary Outcome: Biomarkers of Inflammation-airway XO Activity
Description: To determine whether, compared to baseline, treatment with NOx + CLA can effect airway XO activity determined in endobronchial biopsies
Time Frame: Before treatment at baseline and after treatment at 8 weeks
Population: Data were not collected for this Outcome Measure. The proposed aims could not be addressed with scientific rigor since the number of subjects who completed the study was very low.
Arm/Group | Conjugated Linolenic Acid + NOx
Number analyzed (Participants) | 0

6. Secondary Outcome: Biomarkers of Inflammation-15NO2-cLA
Description: To determine whether, compared to baseline, treatment with NOx + CLA can effect measurement of 15NO2-cLA in urine.
Time Frame: Before treatment at baseline and after treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: nmoles/mg creatinine
Arm/Group | Conjugated Linolenic Acid + NOx
Number analyzed (Participants) | 6
nmoles/mg creatinine | 9.32 (8.9)
Statistical Analysis 1: Comparison: Conjugated Linolenic Acid + NOx; Test type: Other; p <= 0.05, t-test, 1 sided

7. Secondary Outcome: Biomarkers of Inflammation-anion Superoxide
Description: To determine whether, compared to baseline, treatment with NOx + CLA can decrease production of anion superoxide in fresh airway epithelial cells
Time Frame: Before treatment at baseline and after treatment at 8 weeks
Population: as for outcome 5
Arm/Group | Conjugated Linolenic Acid + NOx
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With a Decrease of Inflammation Using Mitochondrial ROS Production
Description: To determine whether, compared to baseline, treatment with NOx + CLA can decrease inflammation using mitochondrial ROS production in fresh and cultured airway epithelial cells.
Time Frame: Before treatment at baseline and after treatment at 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Conjugated Linolenic Acid + NOx
Number analyzed (Participants) | 6
Participants | 0
Statistical Analysis 1: Comparison: Conjugated Linolenic Acid + NOx; Test type: Other; p <= 0.05, t-test, 1 sided

9. Secondary Outcome: Biomarkers of Inflammation- Concentration of NO2-CLA in Plasma
Description: To determine whether, compared to baseline, treatment with NOx + CLA can quantify the concentrations of NO2-cLA in plasma
Time Frame: Before treatment at baseline and after treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: Nanomolar
Arm/Group | Conjugated Linolenic Acid + NOx
Number analyzed (Participants) | 6
Nanomolar | 5.65 (1.48)
Statistical Analysis 1: Comparison: Conjugated Linolenic Acid + NOx; Test type: Other; p <= 0.05, t-test, 1 sided

10. Secondary Outcome: Biomarkers of Inflammation- Concentration of NO2-CLA in Urine
Description: To determine whether, compared to baseline, treatment with NOx + CLA can quantify the concentrations of NO2-cLA in urine
Time Frame: Before treatment at baseline and after treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: nmoles/mg creatinine
Arm/Group | Conjugated Linolenic Acid + NOx
Number analyzed (Participants) | 6
nmoles/mg creatinine | 4.33 (1.8)
Statistical Analysis 1: Comparison: Conjugated Linolenic Acid + NOx; Test type: Other; p <= 0.05, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Before treatment at baseline through completion of treatment at 8 weeks
Description: The occurrence of adverse events was routinely determined through regular investigator/research coordinator assessment.
Arm/Group | Conjugated Linolenic Acid + NOx
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conjugated Linolenic Acid + NOx (N=6)
Headache (General disorders) | 6
Nausea (Gastrointestinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT02433977/Prot_SAP_000.pdf